CLINICAL TRIAL: NCT01977014
Title: NIMS- New Implantable Pump in Pulmonary Arterial Hypertension, a Safety Follow up
Status: Completed | Type: Observational
Sponsor: NordicInfu Care AB (Industry)
Responsible Party: Sponsor
Other Study IDs: NIMS/PAH/LP/001
Record Dates: First submitted 2013-10-22; First posted 2013-11-06 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Hypertension Group 1 and 4 According to Nice Classification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient with LenusPro pump

SUMMARY:
This observational study aims to chart patients which get their prostacyclin treatment via the subcutaneous LenusPro pump. How the surgical procedure is performed and the clinical follow-up of these patients. And by this also charting complications that might occur in relation to treatment.

Participating centres are located in Denmark, Norway and Sweden.

ELIGIBILITY:
Inclusion Criteria:

* The patient should have been diagnosed with Pulmonary Arterial Hypertension
* The patient has received or will receive treatment with the implanted pump LenusPro

Exclusion Criteria:

* The patient is participating in another study which means treatment of the patient no longer follows the normal clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Scandinavia who received a LenusPro pump
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of events reported for the Lenus Pro in a clinical environment. | Up to 3,5 years
Changes in baseline variables during follow-up on quality of life. | Up to 3,5 years
  Patient reported outcome measures, mainly CAMPHOR and SF-36

SECONDARY OUTCOMES:
Description of baseline and follow-up of hemodynamic and functional capacity. | Up to 3,5 years
  Mainly right hearth catheterization, echo and 6MWD data.

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Carlsen, MD, Principal Investigator — Department of Cardiology, Rigshospitalet in Copenhagen; Gerhard Vikstrom, MD, Principal Investigator — Department of Cardiology, Uppsala Akademiska University Hospital; Arne Andreassen, MD, Principal Investigator — Department of Cardiology, Oslo University Hospital
Locations (8):
- Denmark (2):
  - Department of Cardiology, Aarhus University Hospital, Skejby, Aarhus
  - Department of Cardiology Rigshospitalet University Hospital, Copenhagen
- Norway (2):
  - Department of Cardiology Oslo University Hospital, Rikshospitalet, Oslo
  - Department of Cardiology, St Olav University Hospital, Trondheim
- Sweden (4):
  - Department of Cardiology University Hospital in Linköping, Linköping
  - Skane Univerity Hospital, Lund, Lund
  - Karolinska Univerity Hospital, Solna, Stockholm
  - Department of Cardiology Uppsala Akademiska University Hospital, Uppsala